CLINICAL TRIAL: NCT00980109
Title: A Phase IV, Multi-center, Randomized, Partially Double Blinded, Placebo Controlled Study, to Evaluate the Safety of Daily Inhaled Zanamivir 10 mg Versus Placebo and Daily Oral Oseltamivir 75 mg Versus Placebo for Influenza Prophylaxis in Healthy Volunteers for 16 Weeks
Brief Title: Long Term Influenza Prophylaxis With Inhaled Zanamivir or Oral Oseltamivir
Acronym: SEA 004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: The Chancellor, Masters and Scholars of the University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SEA 004; N01AO50042 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Influenza
Keywords: Influenza Prophylaxis; Long Term; Oral Oseltamivir; Inhaled Zanamivir
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Zanamivir; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo oseltamivir (Placebo Comparator): Placebo capsules, one capsule daily for 112 days. The capsule should be administered at approximately the same time each day.
  Interventions: Drug: placebo capsule
- zanamivir for inhalation (Active Comparator): Zanamivir for inhalation, (5 mg per inhalation), two inhalations, once daily using a ROTADISK/DISKHALER for 112 days. The dose should be administered at approximately the same time each day.
  Interventions: Drug: zanamivir for inhalation
- placebo inhalation (Placebo Comparator): Placebo (lactose powder), two inhalations, once daily using a ROTADISK/ DISKHALER for 112 days. The dose should be administered at approximately the same time each day.
  Interventions: Drug: placebo for inhalation
- active oseltamivir (Active Comparator): Oseltamivir capsules (75 mg per capsule), one capsule daily by mouth (PO) for 112 days. The dose should be administered at approximately the same time each day.
  Interventions: Drug: active oseltamivir

INTERVENTIONS:
Drug: active oseltamivir — Oseltamivir capsules (75 mg per capsule), one capsule daily by mouth (PO) for 112 days. The dose should be administered at approximately the same time each day.
  Other Names: Tamiflu
  Arms: active oseltamivir
Drug: placebo capsule — Placebo capsules, one capsule daily for 112 days. The capsule should be administered at approximately the same time each day.
  Arms: placebo oseltamivir
Drug: zanamivir for inhalation — Zanamivir for inhalation, (5 mg per inhalation), two inhalations, once daily using a ROTADISK/DISKHALER for 112 days. The dose should be administered at approximately the same time each day.
  Other Names: Rotadisk/Diskhaler
  Arms: zanamivir for inhalation
Drug: placebo for inhalation — Placebo (lactose powder), two inhalations, once daily using a ROTADISK/ DISKHALER for 112 days. The dose should be administered at approximately the same time each day.
  Arms: placebo inhalation

SUMMARY:
This is a multicenter, randomised, four arms placebo controlled study to evaluate the safety and tolerability of 10 mg inhaled zanamivir once a day and 75 mg oseltamivir capsule orally once a day relative to placebo over 16 weeks (112 days). Enrolled subjects will be randomly assigned to 2:1:2:1 ratio (active oseltamivir: placebo: active zanamivir: placebo) on one of the four study treatment groups.

It is hypothesized that oseltamivir and zanamivir will protect participants from becoming infected with influenza.

DETAILED DESCRIPTION:
We plan to recruit 130 non-pregnant subjects including Health Care Workers, which refer to anyone who works in the hospital, into each active arm and 65 healthy, non-pregnant subjects including Health Care Workers into each placebo arm for a total of 390 study subjects from 4 study sites in Bangkok and Nonthaburi province, Thailand: (i) Faculty of Medicine Siriraj Hospital, (ii) Bamrasnaradura Infectious Diseases Institute, (iii) Chest Disease Institute, and (iv) Hospital for Tropical Diseases.

Randomisation Groups:

Zanamivir for inhalation, (5 mg per inhalation), two inhalations, once daily using a ROTADISK/DISKHALER for 112 days. The dose should be administered at approximately the same time each day.

Placebo (lactose powder), two inhalations, once daily using a ROTADISK/ DISKHALER for 112 days. The dose should be administered at approximately the same time each day.

Oseltamivir capsules (75 mg per capsule), one capsule daily by mouth (PO) for 112 days. The dose should be administered at approximately the same time each day.

Placebo capsules, one capsule daily for 112 days. The capsule should be administered at approximately the same time each day.

Study duration

The study is expected to last up to about 12 months. The study will consist of:

* a screening visit
* 10 study visits: Days 0 , 7 (+2), 14 (+2), 28 (+2), 42 (+2), 56 (+2), 70 (+2), 84 (+2), 98 (+2) and 112 (+2) and
* One follow-up visit on Day 120 (+2)

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:

  1. Healthy male or female aged 20 - 65 years. Healthy determined by the Investigator based on medical history and screening examinations.
  2. Read and understand study related materials intended for subject.
  3. Signed informed consent prior to study participation.
  4. Willingness and ability to comply with the study protocol for the duration of the trial.
  5. Female subject who is of reproductive potential agrees to use an acceptable method of birth control (e.g., intrauterine device, abstinence or hormonal contraceptive drug) throughout the study (D120+2).
  6. For male subject, he must agree to use an acceptable method of birth control (e.g. abstinence or condom) throughout the study (D120+2).

     Exclusion Criteria:
* A subject will not be eligible for inclusion in this study if any of the following apply:

  1. Females who are pregnant, trying to get pregnant or are lactating.
  2. Current or a history of asthma or chronic obstructive pulmonary disease within the last 5 years.
  3. Abnormal pulmonary function test according to The Thoracic Society of Thailand Guidelines for Pulmonary Function Tests: (i) FVC < 80% of the predicted value for age and sex or (ii) FEV1/FVC <70%. (see Appendix 2)
  4. Any other chronic or acute diseases requiring treatment.
  5. An abnormal ECG indicating disease that requires immediate investigation or treatment
  6. An abnormal chest x-ray indicating an active disease process.
  7. A creatinine clearance < 30 mL/min as determined by Cockcroft-Gault equation (see below)
  8. AST or ALT ≥ 1.5 x ULN
  9. Use of a live attenuated influenza vaccine or any anti-influenza drug within 14 days prior to the first dose of study drugs/placebos.
  10. History of alcohol or substance abuse or dependence which in the opinion of the investigator would interfere with subject compliance or safety
  11. Subjects who have a history of allergy to the study drug or drugs of the same class, or a history of severe drug (e.g. toxic epidermal necrolysis) or other allergy (e.g. previous history of anaphylaxis) that, in the opinion of the investigator, contraindicates participation in the trial.
  12. The subject has participated in a clinical trial and has received investigational drugs within 60 days prior to the first dose of study drug.
  13. Subjects who, in the opinion of the investigator, are unlikely to comply fully with study procedures.
  14. History of any mental illness requiring hospitalisation or outpatient psychiatric treatment within the last 12 months
  15. Any suicidal attempt within the previous 5 years.
  16. Screening HADS anxiety or depression score > 8.
  17. Hemoglobin <11g/dL or neutropenia of < 1000 per microlitre or a platelet count of less than 100,000 cells/mm3 Cockroft formula: CrCl (mL/min) = (140 - age) x Wt / 72 x serum creatinine (females x 0.85), age in years, Wt in kg, serum creatinine in mg/dL.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who withdraw from the study because of serious adverse events (SAEs) that are possibly or probably or definitely related to the study drug | 1 year

SECONDARY OUTCOMES:
Proportion of subjects who withdraw from the study because of SAEs unlikely or not related to study drug/placebo | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Bangkok, Bangkoknoi
  - Hospital for Tropical Diseases, Bangkok